CLINICAL TRIAL: NCT01709682
Title: Progression of Atrial Fibrillation After a Failed Initial Ablation Procedure in Patients With Paroxysmal Atrial Fibrillation: A Randomized Comparison of the Drug Therapy Versus Re-Ablation
Brief Title: A Comparison of the Drug Therapy Versus Re-Ablation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAF-DT-RA
Record Dates: First submitted 2012-10-11; First posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Paroxysmal Atrial Fibrillation; Failed First Radiofrequency Ablation Procedure
Keywords: atrial fibrillation; arrhythmias; anti-arrhythmic agents
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Anti-Arrhythmia Agents; Propafenone; Flecainide; Sotalol; Amiodarone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AAD therapy (Active Comparator): Recurrent episodes were pharmacologically managed by conventional AAD therapy (propafenone, flecainide, and/or sotalol as first-line drugs in patients without structural heart disease or amiodarone as a single drug or in combination in patients with structural heart disease or in case of first-line drug failure) according to AF management guidelines.
  Interventions: Drug: Anti-Arrhythmia Agents (propafenone, flecainide, and/or sotalol, or amiodarone); Procedure: ILR implantation
- re-ablation procedure (Active Comparator): Reisolation of the PVs was performed by identifying the breakthrough site on the mapping catheter (NaviStar ThermoCool, Biosense-Webster Inc., Diamond Bar, CA). RF energy was delivered at 43°C, 35 W, 0.5 cm away from the PV ostia at the anterior wall, and was reduced to 43°C, 30 W, 1 cm away from the PV ostia at the posterior wall, with a saline irrigation rate of 17 mL/min. Each lesion was ablated continuously until the local potential amplitude decreased by >80% or RF energy deliveries exceeded 40 s.
  The endpoint of ablation was complete PVI; this was confirmed when Lasso catheter mapping showed the disappearance of all PV potentials or the dissociation of PV potentials from LA activity. Only in patients with induced left atrial flutter, additional RF ablation lines were created by connecting the left inferior PV to the mitral annulus (mitral isthmus) and the roof of the LA between the two superior PVs.
  Interventions: Procedure: re-ablation procedure; Procedure: ILR implantation

INTERVENTIONS:
Drug: Anti-Arrhythmia Agents (propafenone, flecainide, and/or sotalol, or amiodarone) — propafenone, flecainide, and/or sotalol as first-line drugs in patients without structural heart disease or amiodarone as a single drug or in combination in patients with structural heart disease or in case of first-line drug failure
  Arms: AAD therapy
Procedure: re-ablation procedure — Reisolation of the PVs was performed by identifying the breakthrough site on the mapping catheter (NaviStar ThermoCool, Biosense-Webster Inc., Diamond Bar, CA). RF energy was delivered at 43°C, 35 W, 0.5 cm away from the PV ostia at the anterior wall, and was reduced to 43°C, 30 W, 1 cm away from the PV ostia at the posterior wall, with a saline irrigation rate of 17 mL/min. Each lesion was ablated continuously until the local potential amplitude decreased by >80% or RF energy deliveries exceeded 40 s. The endpoint of ablation was complete PVI; this was confirmed when Lasso catheter mapping showed the disappearance of all PV potentials or the dissociation of PV potentials from LA activity.
  Arms: re-ablation procedure
Procedure: ILR implantation — The Reveal XT was implanted in the parasternal area of the chest. The requirement for defining the exact final position was an R-wave amplitude ≥0.4 mV assessed through the Vector Check.
  Patients were provided with the Patient Assistant, a tool that allows each patient to store the ECG through the implanted device during symptoms; data were collected in order to analyze heart rhythm during symptomatic events.

SUMMARY:
The hypothesis of this study was that early re-ablation (test) was superior to AAD therapy (control) in patients with previous failed PVI ablation for paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

* history of symptomatic PAF

Exclusion Criteria:

* congestive heart failure
* LV ejection fraction < 35%
* left atrial diameter > 60 mm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2007-11; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
progression of AF (AF burden progression and persistent AF) | 3 year

SECONDARY OUTCOMES:
recurrence of atrial tachyarrhythmia, including AF and atrial flutter/tachycardia | 3 years
number of further ablation | 3 years
predictors of AF progression | 3 years
  AF burden by ILR monitoring
complications | 3 years
  * tamponade
  * pulmonary vein stenosis
  * atrio-esophora fistula (for re-ablation arm)
  * ventricular arrhythmia
  * symptomatic bradycardia (for AAD arm)

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Derived] Pokushalov E, Romanov A, De Melis M, Artyomenko S, Baranova V, Losik D, Bairamova S, Karaskov A, Mittal S, Steinberg JS. Progression of atrial fibrillation after a failed initial ablation procedure in patients with paroxysmal atrial fibrillation: a randomized comparison of drug therapy versus reablation. Circ Arrhythm Electrophysiol. 2013 Aug;6(4):754-60. doi: 10.1161/CIRCEP.113.000495. Epub 2013 Jun 7. PMID 23748210
- See also: State Research Institute of Circulation Pathology Official Site — http://www.meshalkin.ru/